CLINICAL TRIAL: NCT04836325
Title: Effect of Transcranial Static Magnetic Field Stimulation Over the Primary Motor Cortex in Fibromyalgia Syndrome: A Randomized Controlled Pilot Study
Brief Title: Effect of Transcranial Static Magnetic Field Stimulation in Fibromyalgia Syndrome
Acronym: TSMFS-FMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Seville (Other)
Responsible Party: Principal Investigator, JJ JIMENEZ-REJANO, PhD, University of Seville
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: JJJimenez-Rejano, USeville
Record Dates: First submitted 2021-03-30; First posted 2021-04-08 (Actual); Last update posted 2022-06-08 (Actual); Status verified 2022-06

CONDITIONS: Fibromyalgia
Keywords: transcranial static magnetic field stimulation; fibromyalgia; pain
MeSH Terms: conditions — Fibromyalgia; Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: transcranial static magnetic field stimulation (tSMS) (Experimental): The intervention group will receive a treatment of Transcranial Static Magnetic Field Stimulation (tSMS) in the primary motor cortex with a duration of 30 minutes, 5 times a week, during 4 weeks, for a total of 20 sessions.
  Interventions: Procedure: transcranial static magnetic field stimulation (tSMS)
- Sham transcranial static magnetic field stimulation (Sham Comparator): The placebo group will receive a dummy treatment with a duration of 30 minutes, 5 times a week, during 4 weeks, for a total of 20 sessions.
  Interventions: Procedure: Sham transcranial static magnetic field stimulation

INTERVENTIONS:
Procedure: transcranial static magnetic field stimulation (tSMS) — The intervention group will receive a treatment of tSMS in the primary motor cortex.
  Arms: Experimental: transcranial static magnetic field stimulation (tSMS)
Procedure: Sham transcranial static magnetic field stimulation — The placebo group will receive a dummy treatment
  Arms: Sham transcranial static magnetic field stimulation

SUMMARY:
The main objective is to know if the transcranial static magnetic field stimulation (tSMS) reduces the perception of pain in patients with fibromyalgia and its effect on health-related quality of life. In addition, it will seek to limit the parameters necessary to achieve efficiency with the technique.

DETAILED DESCRIPTION:
Background:

Various non-invasive brain stimulation techniques have been successfully tested in fibromyalgia syndrome (FMS). Transcranial static magnetic field stimulation (tSMS) is a new, portable and inexpensive non invasive brain stimulation (NIBS) technique that has shown security, biological effects, and therapeutical effects in some pathologies. Some studies have studied its effect in pain central processing, our aim is to study its effect on FMS. The safety that tSMS has demonstrated in several clinical trials opens doors to future clinical trials that will extend its clinical utility.

Objectives:

To investigate the effect of tSMS on pain in patients with FMS, using subjective and objective assessment measures. Identify dose response to the treatment to limit the parameters required to achieve effectiveness with the technique.

ELIGIBILITY:
Inclusion Criteria:

* Formal diagnosis of fibromyalgia syndrome (FMS).
* No change in the last 4 weeks on their standard treatment.
* They must have pain for more than 6 months (at least 4 on the VAS scale).
* Score on the fibromyalgia impact questionnaire (FIQ) greater than 39.

Exclusion Criteria:

* Presence of concomitant autoimmune or hematologic diseases.
* Neuropsychiatric disorders.
* Pacemakers or neurostimulators implants.
* Substance abuse or other pathologies that can explain chronic pain.
* Pregnant or lactating women.
* Those who are receiving any other type of physiotherapy treatment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2021-04-19 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Change from Self-reported pain intensity | At the start of the study (at baseline, 0 week), after the 10th session (at the end of the second week), after 20th session (at the end of the fourth week), 1 month from the last session (8th week) and 3 months from the last session (16th week)
  Self-reported pain intensity evaluated by the Visual Analogue Scale (VAS).
Change from Self-reported quality of life | At the start of the study (at baseline, 0 week), after the 10th session (at the end of the second week), after 20th session (at the end of the fourth week), 1 month from the last session (8th week)) and 3 months from the last session (16th week)
  Self-reported quality of life evaluated by the Fibromyalgia Impact Questionnaire (FIQ).

SECONDARY OUTCOMES:
Change from Self-reported catastrophizing | At the start of the study (at baseline, 0 week), after the 10th session (at the end of the second week), after 20th session (at the end of the fourth week), 1 month from the last session (8th week)) and 3 months from the last session (16th week)
  Self-reported catastrophizing evaluated by the Pain Catastrophizing Scale: 13 items, using the 0 (not at all) to 4 (all the time) scale. A total score is yielded (ranging from 0-52), the worse the result the higher the score.
Change from Confidence in the treatment | After the 10th session (at the end of the second week), after 20th session (at the end of the fourth week), 1 month from the last session (8th week)) and 3 months from the last session (16th week)
  Confidence in the treatment evaluated by the Patient Global Impression of Change.
Change from Global health | At the start of the study (at baseline, 0 week), after the 10th session (at the end of the second week), after 20th session (at the end of the fourth week), 1 month from the last session (8th week)) and 3 months from the last session (16th week)
  Self-reported Global health evaluated by the Short form-36 (SF-36).
Change from Cognitive impairment | At the start of the study (at baseline, 0 week), after the 10th session (at the end of the second week), after 20th session (at the end of the fourth week), 1 month from the last session (8th week)) and 3 months from the last session (16th week)
  Cognitive impairment evaluated by the Multidimensional Inventory of Subjective Cognitive Impairment.
Change from Depression | At the start of the study (at baseline, 0 week), after the 10th session (at the end of the second week), after 20th session (at the end of the fourth week), 1 month from the last session (8th week)) and 3 months from the last session (16th week)
  Depression Evaluated by the Hospital Anxiety and Depression Scale: 14 items, 7 for depression and 7 for anxiety. Each item had been answered by the patient on a four-point (0-3) response category so the possible scores ranged from 0 to 21 for anxiety and 0 to 21 for depression, the worse the result the higher the score.
Change from Sleep | At the start of the study (at baseline, 0 week), after the 10th session (at the end of the second week), after 20th session (at the end of the fourth week), 1 month from the last session (8th week)) and 3 months from the last session (16th week)
  Change from Sleep evaluated by the Medical Outcomes Study Sleep Scale:12 Likert-type items with 6 degrees of response (from 1-always to 6-never). For its interpretation, a gross estimate of the amount of sleep is obtained (item 2) and scores in the different subscales. The direct scores are transformed into a scale from 0 to 100, with no cut-off points; the higher the score, the greater the intensity of the concept evaluated.
Change from Physical activity | After the 10th session (at the end of the second week), after 20th session (at the end of the fourth week), 1 month from the last session (8th week) and 3 months from the last session (16th week)
  Change from Physical activity evaluated by the International Physical Activity Questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: JOSE-JESUS JIMENEZ-REJANO, PhD, Study Director — University of Seville
Locations (1):
- Grupo de Investigación Área de Fisioterapia CTS 305 - Universidad de Sevilla, Seville, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Eich W, Bar KJ, Bernateck M, Burgmer M, Dexl C, Petzke F, Sommer C, Winkelmann A, Hauser W. [Definition, classification, clinical diagnosis and prognosis of fibromyalgia syndrome : Updated guidelines 2017 and overview of systematic review articles]. Schmerz. 2017 Jun;31(3):231-238. doi: 10.1007/s00482-017-0200-7. German. PMID 28421273
- [Result] Wolfe F, Walitt B. Culture, science and the changing nature of fibromyalgia. Nat Rev Rheumatol. 2013 Dec;9(12):751-5. doi: 10.1038/nrrheum.2013.96. Epub 2013 Jul 2. PMID 23820862
- [Result] Wolfe F, Clauw DJ, Fitzcharles MA, Goldenberg DL, Katz RS, Mease P, Russell AS, Russell IJ, Winfield JB, Yunus MB. The American College of Rheumatology preliminary diagnostic criteria for fibromyalgia and measurement of symptom severity. Arthritis Care Res (Hoboken). 2010 May;62(5):600-10. doi: 10.1002/acr.20140. PMID 20461783
- [Result] Wolfe F, Clauw DJ, Fitzcharles MA, Goldenberg DL, Hauser W, Katz RS, Mease P, Russell AS, Russell IJ, Winfield JB. Fibromyalgia criteria and severity scales for clinical and epidemiological studies: a modification of the ACR Preliminary Diagnostic Criteria for Fibromyalgia. J Rheumatol. 2011 Jun;38(6):1113-22. doi: 10.3899/jrheum.100594. Epub 2011 Feb 1. PMID 21285161
- [Result] Serra J, Collado A, Sola R, Antonelli F, Torres X, Salgueiro M, Quiles C, Bostock H. Hyperexcitable C nociceptors in fibromyalgia. Ann Neurol. 2014 Feb;75(2):196-208. doi: 10.1002/ana.24065. Epub 2014 Feb 12. PMID 24243538
- [Result] Gentile E, Ricci K, Delussi M, Brighina F, de Tommaso M. Motor Cortex Function in Fibromyalgia: A Study by Functional Near-Infrared Spectroscopy. Pain Res Treat. 2019 Jan 16;2019:2623161. doi: 10.1155/2019/2623161. eCollection 2019. PMID 30792923
- [Result] Di Lazzaro V, Oliviero A, Pilato F, Saturno E, Dileone M, Mazzone P, Insola A, Tonali PA, Rothwell JC. The physiological basis of transcranial motor cortex stimulation in conscious humans. Clin Neurophysiol. 2004 Feb;115(2):255-66. doi: 10.1016/j.clinph.2003.10.009. PMID 14744565
- [Result] Groppa S, Oliviero A, Eisen A, Quartarone A, Cohen LG, Mall V, Kaelin-Lang A, Mima T, Rossi S, Thickbroom GW, Rossini PM, Ziemann U, Valls-Sole J, Siebner HR. A practical guide to diagnostic transcranial magnetic stimulation: report of an IFCN committee. Clin Neurophysiol. 2012 May;123(5):858-82. doi: 10.1016/j.clinph.2012.01.010. Epub 2012 Feb 19. PMID 22349304
- [Result] Lefaucheur JP, Antal A, Ayache SS, Benninger DH, Brunelin J, Cogiamanian F, Cotelli M, De Ridder D, Ferrucci R, Langguth B, Marangolo P, Mylius V, Nitsche MA, Padberg F, Palm U, Poulet E, Priori A, Rossi S, Schecklmann M, Vanneste S, Ziemann U, Garcia-Larrea L, Paulus W. Evidence-based guidelines on the therapeutic use of transcranial direct current stimulation (tDCS). Clin Neurophysiol. 2017 Jan;128(1):56-92. doi: 10.1016/j.clinph.2016.10.087. Epub 2016 Oct 29. PMID 27866120
- [Result] Capone F, Dileone M, Profice P, Pilato F, Musumeci G, Minicuci G, Ranieri F, Cadossi R, Setti S, Tonali PA, Di Lazzaro V. Does exposure to extremely low frequency magnetic fields produce functional changes in human brain? J Neural Transm (Vienna). 2009 Mar;116(3):257-65. doi: 10.1007/s00702-009-0184-2. Epub 2009 Feb 3. PMID 19189041
- [Result] Capone F, Pellegrino G, Motolese F, Rossi M, Musumeci G, Di Lazzaro V. Extremely Low Frequency Magnetic Fields Do Not Affect LTP-Like Plasticity in Healthy Humans. Front Hum Neurosci. 2020 Feb 5;14:14. doi: 10.3389/fnhum.2020.00014. eCollection 2020. PMID 32116603
- [Result] Oliviero A, Mordillo-Mateos L, Arias P, Panyavin I, Foffani G, Aguilar J. Transcranial static magnetic field stimulation of the human motor cortex. J Physiol. 2011 Oct 15;589(Pt 20):4949-58. doi: 10.1113/jphysiol.2011.211953. Epub 2011 Aug 1. PMID 21807616
- [Result] Shibata S, Watanabe T, Yukawa Y, Minakuchi M, Shimomura R, Mima T. Effect of transcranial static magnetic stimulation on intracortical excitability in the contralateral primary motor cortex. Neurosci Lett. 2020 Apr 1;723:134871. doi: 10.1016/j.neulet.2020.134871. Epub 2020 Feb 25. PMID 32109553
- [Result] Oliviero A, Carrasco-Lopez MC, Campolo M, Perez-Borrego YA, Soto-Leon V, Gonzalez-Rosa JJ, Higuero AM, Strange BA, Abad-Rodriguez J, Foffani G. Safety Study of Transcranial Static Magnetic Field Stimulation (tSMS) of the Human Cortex. Brain Stimul. 2015 May-Jun;8(3):481-5. doi: 10.1016/j.brs.2014.12.002. Epub 2014 Dec 11. PMID 25595064
- [Result] Dileone M, Mordillo-Mateos L, Oliviero A, Foffani G. Long-lasting effects of transcranial static magnetic field stimulation on motor cortex excitability. Brain Stimul. 2018 Jul-Aug;11(4):676-688. doi: 10.1016/j.brs.2018.02.005. Epub 2018 Feb 7. PMID 29500043
- [Result] Kirimoto H, Tamaki H, Otsuru N, Yamashiro K, Onishi H, Nojima I, Oliviero A. Transcranial Static Magnetic Field Stimulation over the Primary Motor Cortex Induces Plastic Changes in Cortical Nociceptive Processing. Front Hum Neurosci. 2018 Feb 15;12:63. doi: 10.3389/fnhum.2018.00063. eCollection 2018. PMID 29497371
- [Result] Knijnik LM, Dussan-Sarria JA, Rozisky JR, Torres IL, Brunoni AR, Fregni F, Caumo W. Repetitive Transcranial Magnetic Stimulation for Fibromyalgia: Systematic Review and Meta-Analysis. Pain Pract. 2016 Mar;16(3):294-304. doi: 10.1111/papr.12276. Epub 2015 Jan 12. PMID 25581213
- [Result] Lloyd DM, Wittkopf PG, Arendsen LJ, Jones AKP. Is Transcranial Direct Current Stimulation (tDCS) Effective for the Treatment of Pain in Fibromyalgia? A Systematic Review and Meta-Analysis. J Pain. 2020 Nov-Dec;21(11-12):1085-1100. doi: 10.1016/j.jpain.2020.01.003. Epub 2020 Jan 23. PMID 31982685
- [Result] Paolucci T, Piccinini G, Iosa M, Piermattei C, de Angelis S, Grasso MR, Zangrando F, Saraceni VM. Efficacy of extremely low-frequency magnetic field in fibromyalgia pain: A pilot study. J Rehabil Res Dev. 2016;53(6):1023-1034. doi: 10.1682/JRRD.2015.04.0061. PMID 28475205
- [Result] Kirimoto H, Tamaki H, Matsumoto T, Sugawara K, Suzuki M, Oyama M, Onishi H. Effect of transcranial static magnetic field stimulation over the sensorimotor cortex on somatosensory evoked potentials in humans. Brain Stimul. 2014 Nov-Dec;7(6):836-40. doi: 10.1016/j.brs.2014.09.016. Epub 2014 Sep 30. PMID 25444588
- [Result] Kirimoto H, Asao A, Tamaki H, Onishi H. Non-invasive modulation of somatosensory evoked potentials by the application of static magnetic fields over the primary and supplementary motor cortices. Sci Rep. 2016 Oct 4;6:34509. doi: 10.1038/srep34509. PMID 27698365